CLINICAL TRIAL: NCT04468945
Title: Effects of Mirror Therapy Versus Repetitive Facilitation Exercise on Upper Limb Function in Post-stroke Patient
Brief Title: Mirror Therapy Versus Repetitive Facilitation Exercise on Upper Limb Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00556 Saba Karamat
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Stroke Patient
Keywords: Mirror therapy; Repetitive Facilitation Exercise; stroke; Upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mirror box therapy (Experimental): The objects use for task-specific mirror therapy are duster, glass, the wooden block of different sizes and shapes, beads, coin, paper cards and spongy ball. In all these activities shoulder horizontal flexion-extension, adduction-abduction, elbow flexion-extension, forearm supination-pronation, wrist flexion-extension, finger flexion-extension, abduction, adduction, opposition, are performed automatically.
  Interventions: Other: mirror box therapy
- Repetitive Facilitation Exercise (Experimental): Treatment involved rapid passive stretching of the muscles of the targeted joints in conjunction with tapping and rubbing the skin to assist in the generation of a contraction.Shoulder horizontal flexion-extension , adduction-abduction ,elbow flexion-extension, forearm supination-pronation, wrist flexion-extension, finger flexion-extension, abduction, adduction, opposition, are performed
  Interventions: Other: Repetitive Facilitation Exercise

INTERVENTIONS:
Other: mirror box therapy — * Patients in Task-specific mirror box therapy group will receive therapy for 30 min/day, 3 times/week for 6 weeks.
  * The patient is seated close to a table a mirror (33*35 cm) was placed vertically. The involved hand was placed behind the mirror and uninvolved in front of the mirror.
  * The subject is asked to transfer small cubes from the middle position to the lateral side, placing pegs in holes and taking them out, turning over paper cards, placing steel needles in holes, stacking blocks, and putting glass on a shelf.
  * During the sessions, subjects will be asked to try and do the activity on the unaffected side and asked to do some movement with the paretic hand simultaneously.
  Arms: mirror box therapy
Other: Repetitive Facilitation Exercise — * The patients in the control group will receive Repetitive Facilitation Exercise for 30 min/day, 3 times/week for 6 weeks.
  * Repetitive facilitative techniques were used to elicit movement of the shoulder, elbow, wrist, and fingers in a manner designed to minimize synergistic movements.
  * Participants were directed to concentrate on generating movement on the joint being treated while avoiding contraction of non-targeted muscles.
  * Therapists provided verbal directions with commands such as "bend/straighten" or "one, two, three.
  * Participant efforts were supplemented as necessary to achieve a full range of motion (ROM)
  Arms: Repetitive Facilitation Exercise

SUMMARY:
The objective of the study is to determine the effects of Mirror therapy on upper limb function in a post-stroke patient, To determine the effects of Repetitive Facilitation Exercise on upper limb function in a post-stroke patient and To compare the effects of Mirror therapy versus Repetitive Facilitation Exercise on upper limb function in the post-stroke patient. Study Design is Randomized control trial with a sample size of 50 participants. Sampling Technique used is Non-probability purposive assessor-blinded sampling technique and randomization through sealed envelope method Duration of study was 6 months.Study Setting of Railway general hospital. Inclusion criteria had Hemiparetic patient, Sub-acute and chronic stroke patients, First-ever stroke patient, Age: 40-60, Gender: both male and female, MMSE >24, Modified Ashworth scale <3, Stable patient (Good sitting balance ) and No visual-spatial hemineglect. Exclusion criteria of Unstable patient, Uncooperative patient, Orthopedic deformity, Aphasia, Visual infection and joint pain (shoulder, elbow, wrist, hip, knee, ankle)

DETAILED DESCRIPTION:
Stroke is classically characterized as a neurological deficit attributed to an acute focal injury of the central nervous system by a vascular cause, including cerebral infarction, intracerebral haemorrhage, and subarachnoid haemorrhage, and is a major cause of disability and death worldwide. Stroke is the second leading cause of death and the third leading cause of disability. Stroke, the sudden death of some brain cells due to lack of oxygen when the blood flow to the brain is lost by blockage or rupture of an artery to the brain, is also a leading cause of dementia and depression. Stroke kills about 140,000 Americans each year that's 1 out of every 20 deaths. In Pakistan, the stroke incidence of 95 per 100,000 persons per year for the following Years 2000 to 2016, with the highest incidence being 584,000 of 650,000, noted among individuals aged 75 to 85. The paretic upper limb is a common and undesirable consequence of stroke that increases activity limitation. A number of interventions have been published evaluating the effect of various rehabilitation methods improving upper extremity control and functioning. Mirror therapy is a relatively new therapeutic intervention which is simple, inexpensive and most importantly patient-directed treatment that focuses on moving the unimpaired limb. It was first introduced by Ramachandran and Roger Ramachandran to treat phantom limb pain after amputation.The principle of mirror therapy (MT) is use of a mirror to create reflective illusion of an affected limb in order to trick the brain into thinking movement has occurred without pain. It involves placing the affected limb behind a mirror, which is sited to the reflection of the opposing limb appears in placing of the hidden limb. During performing the tasks with the unaffected hand, the participants were instructed to move their affected arm synchronically in the same way while viewing the mirror during the practices with the unaffected arm, the participants were instructed to move their affected arm synchronically while viewing the mirror. Repetitive facilitative exercise (RFE), a combination of high repetition rate and neuro facilitation, is a recently developed approach to the rehabilitation of stroke-related limb impairment. The RFE sessions used a novel facilitation technique to elicit movements of the shoulder, elbow and each finger isolated from synergy and give sufficient physical stimulation, such as by the stretch reflex or skin-muscle reflex that is elicited immediately before or at the same time as when the patient makes an effort to move his hemiplegic hand or finger. Functional recovery of the hemiplegic upper limb and hand might depend on the repetition of voluntary movements elicited by the RFEs, especially when they are influenced by a synergistic pattern. Principles for selection and treatment included the following: (1) an emphasis on the proximal musculature, given its role in stabilizing distal movements, gradual increases in movement difficulty with a goal of maintaining movement purity and avoiding synergy; and consideration of the importance/nature of the movement (eg, the first and second fingers were trained separately and the third and fourth together to facilitate the acquisition of pinch. This aim of the study is to improve the function of the upper limb in post-stroke hemiparesis patient. Repetitive Facilitation exercise has proved beneficial effects for improving upper limb function on stroke patients. There is also different opinion about the effectiveness of Mirror therapy on upper limb function. So the purpose of my study is to investigate whether Mirror Therapy or Repetitive Facilitation exercise is more effective in improving upper limb function in Stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparetic patient
* Sub-acute and chronic stroke patients
* First-ever stroke patient
* Age: 40-60
* Gender: both male and female
* MMSE >24
* Modified Ashworth scale <3
* Stable patient (Good sitting balance )
* No visual-spatial hemineglect.

Exclusion Criteria:

* Unstable patient
* Uncooperative patient
* Orthopaedic deformity
* Aphasia
* Visual infection
* Joint pain (shoulder, elbow, wrist, hip, knee, ankle)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Fugal Meyer scale | From baseline to 6th week
  Fugl Meyer assessment tool is used for the evaluation of recovery extent in post stroke patients. It consists of 226 total points and is divided in 5 major domains including sensory function, motor function, joint range of motion, balance and pain each domain contain multiple sub items. Scoring is being recorded on a (3-points ordinal scale) . upper limb total score is 66. Fugyl Meyer is also a reliable and highly valid tool with ICC=0.96 and internal consistency is 94.7%.
Wolf motor scale | From baseline to 6th week
  The Wolf motor scale is considered as numerical catalogue for the assessment of upper extremity motor function. Motor skills of patients are assessed through time and well designed, practical and functional tasks. Total 15 task has been performed. the minimum value for each task is 1 and maximum value is 3. increased value shows improvement.This is also a reliable tool for upper limb motor function with fair inter rater reliability as the value of ICC=0.97-0.99 and internal consistency is 92.4%.
Upper extremity functional index | From baseline to 6th week
  Upper extremity functional index is use for outcome measure in stroke patient. It consist of 20-item questionnaire and each item has 5 point ordinal scale The total sum of all item the final score is 80 point. The reliability of upper extremity functional index is (ICC=0.94)
Brunnstrom scale | From baseline to 6th week
  Brunnstrom recovery scale is use for motor recovery in stroke patient .It consist of 7-stages, 1=Flaccid Paralysis,2=Spasticity,3=Spasticity is marked ,4=Spasticity decreased,5= Spasticity wanes,6= Coordination and pattern of movement can be near normal ,7=Normal The inter-rater reliability if burnnstrom recovery scale is (ICC 0.89-0.98) for arm and (ICC 0.69-0.92)for hand.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Background] Owolabi MO, Akarolo-Anthony S, Akinyemi R, Arnett D, Gebregziabher M, Jenkins C, Tiwari H, Arulogun O, Akpalu A, Sarfo FS, Obiako R, Owolabi L, Sagoe K, Melikam S, Adeoye AM, Lackland D, Ovbiagele B; Members of the H3Africa Consortium. The burden of stroke in Africa: a glance at the present and a glimpse into the future. Cardiovasc J Afr. 2015 Mar-Apr;26(2 Suppl 1):S27-38. doi: 10.5830/CVJA-2015-038. PMID 25962945
- [Background] Yang Q, Tong X, Schieb L, Vaughan A, Gillespie C, Wiltz JL, King SC, Odom E, Merritt R, Hong Y, George MG. Vital Signs: Recent Trends in Stroke Death Rates - United States, 2000-2015. MMWR Morb Mortal Wkly Rep. 2017 Sep 8;66(35):933-939. doi: 10.15585/mmwr.mm6635e1. PMID 28880858
- [Background] Scheid A, Choppin PW. Two disulfide-linked polypeptide chains constitute the active F protein of paramyxoviruses. Virology. 1977 Jul 1;80(1):54-66. doi: 10.1016/0042-6822(77)90380-4. No abstract available. PMID 195398
- [Background] Shimodozono M, Noma T, Nomoto Y, Hisamatsu N, Kamada K, Miyata R, Matsumoto S, Ogata A, Etoh S, Basford JR, Kawahira K. Benefits of a repetitive facilitative exercise program for the upper paretic extremity after subacute stroke: a randomized controlled trial. Neurorehabil Neural Repair. 2013 May;27(4):296-305. doi: 10.1177/1545968312465896. Epub 2012 Dec 3. PMID 23213077
- [Background] Riggs BL, Jowsey J, Kelly PJ, Arnaud CD. Role of hormonal factors in the pathogenesis of postmenopausal osteoporosis. Isr J Med Sci. 1976 Jul;12(7):615-9. PMID 972016